CLINICAL TRIAL: NCT04869696
Title: Science of Skin: Medical Adhesive Repeat Application Study #2
Brief Title: Medical Adhesive Repeat Application Study
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: EM-05-014952
Record Dates: First submitted 2021-04-08; First posted 2021-05-03 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Skin stripping; TEWL

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tape removed from the skin of subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with tape samples: each subject had 8 types of tape samples applied on their arms

SUMMARY:
This study is to determine the relative effects imparted by different medical tapes to skin when comparing normal skin to skin after ten repeated tape applications and removals.

DETAILED DESCRIPTION:
This study is to evaluate changes to skin after repeated tape stripping on volar forearm with various medical tapes. Assessments of effects to skin include corneocytes, total protein (BCA), Trans-Epidermal Water Loss (TEWL), and cytokine analysis.

The Study will involve the application of eight (8) test articles. In each case, the test articles will be applied to eight (8) sites on the healthy Subject's left and right volar forearms (four [4] sites on the left, and four [4] sites on the right) in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ages 18-65 years.
2. Has sufficient area to fit five (5)1 inch by 2.5-inch sites on each volar forearm.
3. Agrees to have five (5) 1 inch by 2.5-inch test sites marked on each volar forearm with a non-toxic permanent marker (Sharpie).
4. Agrees to stop the use of all topical products (lotions, creams, oils, sunscreen, bug spray, etc.) on their volar forearms 3 days prior to the start of the study.
5. Agrees to not shower within 24 hours of their D1 visit.
6. Agrees to not wash volar forearms when washing hands within 24 hours of their D1 visit.
7. Agrees to refrain from exercising or drinking hot beverages or cold/iced coffee or tea (caffeinated or energy drinks) during the 2 hours prior to their D1 visit.
8. Agrees that if the study personnel feel that they have excessive hair on their volar forearm test sites that the hair may be clipped at the D1 visit.
9. Agrees to wear or be willing to change into a short-sleeved shirt or a shirt with sleeves that can be pulled or rolled above the elbows to each visit.
10. Able to read, understand, and sign the Informed Consent Form (ICF).
11. Willing and able to follow all study requirements and restrictions

Exclusion Criteria:

1. If female, is pregnant, nursing, or planning a pregnancy during the study as determined by interview.
2. If female, is currently experiencing hot flashes (this affects the measurements) or has increased localized or generalized sweating (hyperhidrosis).
3. Is a smoker.
4. Has a history of lightening or darkening of the skin due to tape application and removal.
5. Has diabetes Type 1 or Type 2.
6. Has a current skin condition on the volar forearms (e.g., psoriasis, eczema, atopic dermatitis, etc., or active cancer) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
7. Is currently taking, or in the past 2 weeks has taken any anti-inflammatory drug (e.g., aspirin, ibuprofen, Celebrex [COX-2 inhibitor], corticosteroids), immunosuppressive drugs, or antihistamine medications.
8. Is currently applying, or in the past 2 weeks has applied topical drugs to the volar forearm test sites.
9. Has any medical condition that, in the Investigator's judgment, makes the Subject ineligible or places the Subject at undue risk.
10. Is currently participating in any clinical testing, including other studies being conducted at Dermico LLC.
11. Has damaged skin in or around the test sites, which includes sunburn, extremely deep tans, uneven skin tones, tattoos, scars, excessive hair that they are not willing to have clipped, numerous freckles, blemishes, or other disfiguration of the test sites.
12. Has a confirmed allergy or sensitivity to adhesives.
13. Has a history of a confirmed or suspected COVID-19 infection within 30 days prior to the study visit.
14. Has had contact with a COVID-19-infected person or persons within 14 days prior to the study visit.
15. Individual or a member of the individual's household has traveled internationally within 14 days prior to the study visit.
16. Has experienced any of the following self-reported symptoms of COVID-19 within 2 weeks prior to the study visit:

    * Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomachaches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, or chest pain/tightness.
    * Temperature ≥ 100. 4o F, measured

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will consist of men and women aged 18 to 65 years old, Fitzpatrick Skin Type I-VI. Candidates will be recruited from a pool of healthy men and women who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
Chang in TEWL from skin after repeated tape stripping | Immediately after 10 times of repeated tape application and removal
  Measure change in Transepidermal Water Loss (TEWL) from baseline to Tape 10 after repeated tape applications and removals. Baseline TEWL will be measured on another non-taped site.
Changes to skin after repeated tape stripping (total protein) | After the removal of Tape 1 and after the removal of Tape 10
  Analysis of total protein (BCA) in the skin cells removed by tape samples after repeated tape application and removal. The 1st tape and the 10th tape will be collected for analysis.
Changes to skin after repeated tape stripping (corneocytes) | After the removal of Tape 1 and after the removal of Tape 10
  Analysis of percentage area coverage of corneocytes on the tape samples removed from skin. The 1st tape and the 10th tape will be collected for analysis.
Changes to skin after repeated tape stripping (Cytokine) | Immediately after TEWL measurement is completed on each test site
  Analysis of cytokine in skin cells removed by tape samples after repeated tape application and removal. Cytokine tape collection will take place after the TEWL measurement is completed on each test site. Control cytokine tape will be collected from another non-taped site.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Grove, Principal Investigator — Dermico
Locations (1):
- Dermico, Broomall, Pennsylvania, United States